CLINICAL TRIAL: NCT06637800
Title: Prospective, Open-label Study of Seraph 100 in Patients With Prolonged COVID (PC)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ExThera Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLC01 Prolonged COVID
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Masking Description: Unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Seraph® 100 Microbind® Affinity Blood Filter (Seraph 100) is a single use (Experimental): The Seraph® 100 Microbind® Affinity Blood Filter (Seraph 100) is a single use, disposable column packed with ultra-high molecular weight polyethylene (UHMWPE) beads. These beads have been modified to contain endpoint-attached heparin on the surface, thus forming a new chemical entity, the polymer now containing material of animal origin (porcine mucosa). The devices are sterilized using a standard ethylene oxide (EtO) cycle, following ISO 11135:2014.
  Interventions: Device: Seraph® 100 Microbind® Affinity Blood Filter (Seraph 100)

INTERVENTIONS:
Device: Seraph® 100 Microbind® Affinity Blood Filter (Seraph 100) — The Seraph 100 is part of the Seraph platform technology that was developed as an extracorporeal broad-spectrum sorbent hemoperfusion device for reduction of pathogens, bacteria, viruses, fungus, and other sepsis mediators from the bloodstream. In addition, it has been demonstrated that Seraph 100 is also capable of removing circulating tumor cells from the whole blood.

SUMMARY:
This study will use a prospective, open, single-arm design, in which a group of 100 patients with a diagnosis of prolonged COVID, previously selected according to inclusion and exclusion criteria, and who have undergone informed consent process and have signed the informed consent form, undergo two hemoperfusion procedures with the Seraph 100 filter, on consecutive days. They are then evaluated at day 3 and 4 weeks, to complete the safety and effectiveness assessment.

DETAILED DESCRIPTION:
This will be a prospective, open-label, single-arm, pilot study, in which a group of 100 PC patients will undergo two hemoperfusion procedures, to verify the safety and preliminary efficacy of the Seraph 100 device. Eligible patients will be invited to participate and once they sign the Informed Consent (IC) they will undergo two hemoperfusion procedures, on consecutive days, of -4 hours duration each time, using a multicomponent apheresis machine with the Seraph 100 filter. Patients will be followed for a total of 30 days, to monitor the presence of AEs (safety) and possible changes in clinical outcomes (preliminary efficacy).

ELIGIBILITY:
Inclusion Criteria:

Subjects will be considered eligible for participation in the study if they meet all the following inclusion criteria:

1. Adult patients age of 18-85 (had 18th birthday but did not have 85th birthday).
2. History of COVID 19 infection established by positive polymerase chain reaction (PCR) test or by compatible clinical testing (e.g. rapid antigen, serum testing, or other relevant clinical documentation).
3. Persistent symptoms for 12 or more weeks after acute COVID 19 infection including fatigue and one or more of the following: myalgia or generalized aches and pains; joint pain; dizziness or unsteadiness; cognitive dysfunction (mental fog).
4. Patient (legally designated representative) has completed the Informed Consent process prior to enrollment into this study.
5. Patient (legally designated representative) is willing to comply with the study protocol -

Exclusion Criteria:

Subjects meeting any of the following criteria will not be recruited for the study:

1. History of heparin allergy.
2. History of heparin-induced thrombocytopenia.
3. Pregnancy or breastfeeding.
4. Life expectancy is less than 30 days.
5. The patient is currently enrolled in another drug or device trial. Patients who cannot tolerate placement of double-lumen catheter.
6. Unable to obtain informed consent from either patient or legally authorized representative (LAR)Any subject who, in the investigator's judgment, is considered unsuitable for participation in this trial.

After verification of eligibility and signature of consent:

1. The patient must be able to perform a hemoperfusion procedure with an apheresis machine.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of Technical Procedure Success | Procedure Stop Time
  Procedural Success is defined as:
  1. Device use as originally intended, and
  2. No device procedure related serious adverse events (SAEs)
Assessment of Device Success | 3, 7 and 28 days
  Seraph 100 Device Success

CONTACTS AND LOCATIONS:
Overall Officials: Mink Chawla, M.D., Principal Investigator — ExThera Medical Corporation
Locations (1):
- Hospital Angeles Tijuana, Tijuana, Mexico

IPD SHARING:
Plan to Share IPD: No
Following completion of the study, results of this research will be in a scientific journal. Data will be available immediately following publication, with no end date, with data sharing at the discretion of the Sponsor.